CLINICAL TRIAL: NCT03816696
Title: An Open-Label Two-way Interaction Clinical Trial to Evaluate the Pharmacokinetic Interactions Between GSK3640254 and Dolutegravir in Healthy Subjects
Brief Title: Study to Evaluate the Pharmacokinetic (PK) Interactions Between GSK3640254 and Dolutegravir (DTG)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 209712
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-02

CONDITIONS: HIV Infections
Keywords: GSK3640254, dolutegravir, healthy subjects, two-way interaction, HIV
MeSH Terms: conditions — HIV Infections | interventions — GSK3640254

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DTG followed by GSK3640254 followed by DTG+GSK3640254 (Experimental): Subjects will receive DTG 50 mg QD on Days 1 through 5 in Period 1 followed by a wash-out period of 4 days. Subjects will then receive GSK3640254 200 mg QD on Days 1 through 7 in Period 2 followed by co-administration of DTG 50 mg QD with GSK3640254 200 mg QD on Days 1 through 7 in Period 3.
  Interventions: Drug: GSK3640254; Drug: DTG

INTERVENTIONS:
Drug: GSK3640254 — GSK3640254 will be available as 100 mg capsules. Subjects will be administered GSK3640254 200 mg QD via the oral route.
Drug: DTG — DTG will be available as 50 mg tablets. Subjects will be administered DTG 50 mg QD via the oral route.

SUMMARY:
This is an open-label, single-sequence, two-way drug interaction study to investigate the PK, safety and tolerability of GSK3640254 and DTG when administered alone or in combination in healthy subjects. Treatment of human immunodeficiency virus (HIV) infection frequently involves combination therapy. Data from this study will contribute to dosing recommendations when GSK3640254 and DTG are given in combination. The study will consist of a Screening period and 3 sequential treatment periods. Subjects will be administered DTG 50 milligrams (mg) once daily (QD) in Period 1 followed by GSK3640254 200 mg QD in Period 2. There will be a washout period of 4 days between Periods 1 and 2. In Period 3, subjects will be co-administered DTG 50 mg QD and GSK3640254 200 mg QD. The total duration of the study will be approximately 55 days, including Screening.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Subjects who are healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring (history and ECG).
* Body weight >=50 kilograms (kg) (110 pounds [lbs]) for men and >=45.0 kg (99 lbs) for women and body mass index within the range 18.5 to 31.0 kilograms per square meter (kg/m^2) (inclusive).
* Male or female subjects can participate. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and not a woman of childbearing potential (WOCBP).
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and protocol.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A pre-existing condition interfering with normal gastrointestinal (GI) anatomy or motility (e.g., gastroesophageal reflux disease, gastric ulcers, gastritis), hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs or render the subject unable to take oral study intervention.
* Any history of significant underlying psychiatric disorder, including but not limited to schizophrenia, bipolar disorder with or without psychotic symptoms, other psychotic disorders, or schizotypal (personality) disorder.
* Any history of major depressive disorder with or without suicidal features, or anxiety disorders, that required medical intervention (pharmacologic or not) such as hospitalization or other inpatient treatment and/or chronic (>6 months) outpatient treatment. Subjects with other conditions such as adjustment disorder or dysthymia that have required shorter term medical therapy (<6 months) without inpatient treatment and are currently well-controlled clinically or resolved may be considered for entry after discussion and agreement with the ViiV Medical Monitor.
* Any pre-existing physical or other psychiatric condition (including alcohol or drug abuse), which, in the opinion of the investigator (with or without psychiatric evaluation), could interfere with the subject's ability to comply with the dosing schedule and protocol evaluations or which might compromise the safety of the subject.
* Medical history of cardiac arrhythmias or cardiac disease or a family or personal history of long QT syndrome.
* Presence of Hepatitis B surface antigen (HBsAg) at Screening or within 3 months prior to starting study intervention.
* Positive Hepatitis C antibody test result at Screening or within 3 months prior to starting study intervention and positive on reflex to Hepatitis C ribonucleic acid (RNA).
* Positive HIV-1 and -2 antigen/antibody immunoassay at Screening.
* ALT >1.5 times upper limit of normal (ULN). A single repeat of ALT is allowed within a single screening period to determine eligibility.
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Any acute laboratory abnormality at Screening which, in the opinion of the investigator, should preclude participation in the study of an investigational compound.
* Any Grade 2 to 4 laboratory abnormality at Screening, with the exception of creatine phosphokinase (CPK) and lipid abnormalities (e.g., total cholesterol, triglycerides), and ALT (described above), will exclude a subject from the study unless the investigator can provide a compelling explanation for the laboratory results and has the assent of the sponsor. A single repeat of any laboratory abnormality is allowed within a single screening period to determine eligibility.
* A positive test result for drugs of abuse (including marijuana), alcohol, or cotinine (indicating active current smoking) at Screening or before the first dose of study intervention.
* Unable to refrain from the use of prescription or non-prescription drugs including vitamins, herbal and dietary supplements (including St John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication and for the duration of the study.
* Treatment with any vaccine within 30 days prior to receiving study intervention.
* Unwillingness to abstain from excessive consumption of any food or drink containing grapefruit and grapefruit juice, Seville oranges, blood oranges, or pomelos or their fruit juices within 7 days prior to the first dose of study intervention(s) until the end of the study.
* Participation in another concurrent clinical study or prior clinical study (with the exception of imaging trials) prior to the first dosing day in the current study: 30 days, 5 half-lives, or twice the duration of the biological effect of the study intervention (whichever is longer).
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliter (mL) within 56 days.
* Any positive (abnormal) response confirmed by the investigator on a screening clinician- or qualified designee-administered Columbia Suicide Severity Rating Scale (C-SSRS).
* Any significant arrhythmia or ECG finding (e.g., prior myocardial infarction, sinoatrial pauses, bundle branch block, or conduction abnormality) which, in the opinion of the investigator or ViiV Healthcare (VH)/GlaxoSmithKline (GSK) Medical Monitor, will interfere with the safety for the individual subject.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Heart rate (males: <45 or >100 beats per minute [bpm] and females: <50 or >100 bpm); PR interval (<120 or >200 milliseconds [msec]); QRS duration (<70 or >110 msec); QTcF interval (males: >450 msec and females: >470 msec).
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 units. One unit is equivalent to 8 grams of alcohol: a half-pint (equivalent to 240 mL) of beer, 1 glass (125 mL) of wine, or 1 (25 mL) measure of spirits.
* Regular use of tobacco- or nicotine-containing products within 3 months prior to Screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Pene Dumitrescu T, Joshi SR, Xu J, Greene TJ, Johnson M, Butcher L, Zimmerman E, Webster L, Pham TT, Lataillade M, Min S. Phase I evaluation of pharmacokinetics and tolerability of the HIV-1 maturation inhibitor GSK3640254 and dolutegravir in healthy adults. Br J Clin Pharmacol. 2021 Sep;87(9):3501-3507. doi: 10.1111/bcp.14759. Epub 2021 Mar 4. PMID 33533507

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, fixed-sequence, two-way drug interaction and 3-period study. Participants received treatment A- dolutegravir 50 milligram (mg) in Period 1; treatment B- GSK3640254 200 mg in Period 2 and treatment C- dolutegravir 50 mg and GSK3640254 200 mg in Period 3.
Pre-assignment Details: A total of 30 participants were screened, of which 14 were screening failures. Hence, 16 participants were enrolled in this study. This study was conducted at a single center in the United States.
Groups:
- Dolutegravir/GSK3640254/Dolutegravir+GSK3640254: Participants received treatment A- dolutegravir 50 mg, tablets, orally, once daily on Days 1 to 5 in Period 1; followed by washout period of 4 days between last dose of study treatment A in Period 1 and initiation of study treatment B in Period 2; followed by treatment B- GSK3640254 200 mg, capsules, orally, once daily on Days 1 to 7 in Period 2; further followed by treatment C- dolutegravir 50 mg, tablets, orally, once daily along with GSK3640254 200 mg, capsules, orally, once daily on Days 1 to 7 in Period 3.
Period: Period 1 (Up to Day 5)
Arm/Group | Dolutegravir/GSK3640254/Dolutegravir+GSK3640254
Started | 16
Completed | 16
Not Completed | 0
Period: Wash Out Period (Days 6 to 9)
Arm/Group | Dolutegravir/GSK3640254/Dolutegravir+GSK3640254
Started | 16
Completed | 16
Not Completed | 0
Period: Period 2 (Up to Day 7)
Arm/Group | Dolutegravir/GSK3640254/Dolutegravir+GSK3640254
Started | 16
Completed | 16
Not Completed | 0
Period: Period 3 (Up to Day 11)
Arm/Group | Dolutegravir/GSK3640254/Dolutegravir+GSK3640254
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dolutegravir/GSK3640254/Dolutegravir+GSK3640254
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.7 (10.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 1
  Asian - South East Asian Heritage | 1
  Black or African American | 3
  White - White/Caucasian/European Heritage | 11

OUTCOME MEASURES:

1. Primary Outcome: Period 1: Area Under the Plasma Concentration-time Curve From Time 0 to the End of the Dosing (AUC[0 to Tau]) of Dolutegravir for Dolutegravir Arm
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of dolutegravir. The pharmacokinetic parameters were calculated by standard non-compartmental analysis. Pharmacokinetic Parameter Population consisted of all participants who underwent plasma pharmacokinetic sampling and had evaluable pharmacokinetic parameters estimated.
Time Frame: Day 5: Pre-dose, 1, 1.5, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* nanogram per milliliter
Groups:
- Dolutegravir 50 mg: In Period 1, participants received dolutegravir 50 mg, tablets, orally (treatment A) once daily on Days 1 through 5 followed by a wash-out period of 4 days. A wash out period was maintained between the last dose of study treatment A in Period 1 and initiation of study treatment B in Period 2.
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Hours* nanogram per milliliter | 64627.8 (20.1)

2. Primary Outcome: Period 3: AUC(0 to Tau) of Dolutegravir for Dolutegravir + GSK3640254 Arm
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of dolutegravir. The pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: Day 7: Pre-dose, 1, 1.5, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* nanogram per milliliter
Groups:
- Dolutegravir 50 mg + GSK3640254 200 mg: In Period 3, participants co-administered dolutegravir 50 mg, tablets, orally, once daily along with GSK3640254 200 mg, capsules, orally (treatment C), once daily on Days 1 through 7. Participants were followed up for 4 days after last dose of study treatment.
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Hours* nanogram per milliliter | 75860.5 (22.7)

3. Primary Outcome: Period 1: Maximum Observed Concentration (Cmax) of Dolutegravir for Dolutegravir Arm
Description: as for outcome 2
Time Frame: Day 5: Pre-dose, 1, 1.5, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Nanogram per milliliter | 4962 (16.5)

4. Primary Outcome: Period 3: Cmax of Dolutegravir for Dolutegravir + GSK3640254 Arm
Description: as for outcome 2
Time Frame: Day 7: Pre-dose, 1, 1.5, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Nanogram per milliliter | 5408 (17.2)

5. Primary Outcome: Period 1: Plasma Concentration at the End of the Dosing Interval (Ctau) of Dolutegravir for Dolutegravir Arm
Description: as for outcome 2
Time Frame: Day 5: Pre-dose, 1, 1.5, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Nanogram per milliliter | 1373 (30.6)

6. Primary Outcome: Period 3: Ctau of Dolutegravir for Dolutegravir + GSK3640254 Arm
Description: as for outcome 2
Time Frame: Day 7: Pre-dose, 1, 1.5, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Nanogram per milliliter | 1696 (31.1)

7. Primary Outcome: Period 2: AUC(0 to Tau) of GSK3640254 for GSK3640254 Arm
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of GSK3640254. The pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: Day 7: Pre-dose, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* microgram per milliliter
Groups:
- GSK3640254 200 mg: In Period 2, participants received GSK3640254 200 mg, capsules, orally (treatment B) once daily on Days 1 through 7.
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Hours* microgram per milliliter | 26.72 (32.3)

8. Primary Outcome: Period 3: AUC(0 to Tau) of GSK3640254 for Dolutegravir + GSK3640254 Arm
Description: as for outcome 7
Time Frame: Day 7: Pre-dose, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* microgram per milliliter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Hours* microgram per milliliter | 27.84 (30.1)

9. Primary Outcome: Period 2: Cmax of GSK3640254 for GSK3640254 Arm
Description: as for outcome 7
Time Frame: Day 7: Pre-dose, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Microgram per milliliter | 1.676 (26.4)

10. Primary Outcome: Period 3: Cmax of GSK3640254 for Dolutegravir + GSK3640254 Arm
Description: as for outcome 7
Time Frame: Day 7: Pre-dose, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Microgram per milliliter | 1.662 (26.8)

11. Primary Outcome: Period 2: Ctau of GSK3640254 for GSK3640254 Arm
Description: as for outcome 7
Time Frame: Day 7: Pre-dose, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Microgram per milliliter | 0.8583 (38.3)

12. Primary Outcome: Period 3: Ctau of GSK3640254 for Dolutegravir + GSK3640254 Arm
Description: as for outcome 7
Time Frame: Day 7: Pre-dose, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Microgram per milliliter | 0.8549 (34.1)

13. Secondary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; and other important medical events which may require medical or surgical intervention. Safety Population consisted of all participants who received at least 1 dose of study medication.
Time Frame: Up to Day 27
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir 50 mg | GSK3640254 200 mg | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16 | 16 | 16
Participants
  Non-SAEs | 1 | 3 | 2
  SAEs | 0 | 0 | 0

14. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelet Count
Description: Blood samples were collected to analyze the hematology parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelet count. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day -1) and at Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
10^9 cells per liter
  Basophils | -0.003 (0.0124)
  Eosinophils | 0.046 (0.1198)
  Lymphocytes | 0.013 (0.3793)
  Monocytes | -0.020 (0.0829)
  Neutrophils | -0.217 (0.6421)
  Platelet count | -6.5 (21.73)

15. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelet Count
Description: Blood samples were collected to analyze the hematology parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelet count. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 1 Day 9) and at Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
10^9 cells per liter
  Basophils | -0.006 (0.0089)
  Eosinophils | -0.026 (0.0810)
  Lymphocytes | -0.154 (0.2718)
  Monocytes | -0.024 (0.0701)
  Neutrophils | -0.160 (0.3762)
  Platelet count | -6.0 (30.58)

16. Secondary Outcome: Period 3: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelet Count
Description: Blood samples were collected to analyze the hematology parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelet count. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 2 Day 7) and at Days 4, 7 and 10
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
10^9 cells per liter
  Day 4: Basophils, n=16 | 0.003 (0.0101)
  Day 7: Basophils, n=16 | 0.007 (0.0135)
  Day 10: Basophils, n=16 | 0.003 (0.0144)
  Day 4: Eosinophils, n=16 | -0.001 (0.0448)
  Day 7: Eosinophils, n=16 | 0.004 (0.0846)
  Day 10: Eosinophils, n=16 | -0.036 (0.0468)
  Day 4: Lymphocytes, n=16 | -0.130 (0.2931)
  Day 7: Lymphocytes, n=16 | -0.033 (0.3260)
  Day 10: Lymphocytes, n=16 | -0.117 (0.2628)
  Day 4: Monocytes, n=16 | 0.049 (0.1627)
  Day 7: Monocytes, n=16 | 0.003 (0.0850)
  Day 10: Monocytes, n=16 | -0.018 (0.0693)
  Day 4: Neutrophils, n=16 | 0.443 (1.5098)
  Day 7: Neutrophils, n=16 | 0.076 (0.5969)
  Day 10: Neutrophils, n=16 | 0.204 (0.5116)
  Day 4: Platelet count, n=16 | -4.9 (11.08)
  Day 7: Platelet count, n=15: number analyzed (Participants) | 15
  Day 7: Platelet count, n=15 | -11.5 (12.03)
  Day 10: Platelet count, n=16 | -5.9 (16.50)

17. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day -1) and at Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Grams per liter | 4.4 (5.97)

18. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 1 Day 9) and at Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Grams per liter | 0.1 (2.53)

19. Secondary Outcome: Period 3: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 2 Day 7) and at Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Grams per liter
  Day 4 | 3.3 (3.00)
  Day 7 | 0.6 (3.50)
  Day 10 | 1.2 (3.69)

20. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day -1) and at Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Proportion of red blood cells in blood | 0.0178 (0.01988)

21. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 1 Day 9) and at Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Proportion of red blood cells in blood | -0.0013 (0.00948)

22. Secondary Outcome: Period 3: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 2 Day 7) and at Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Proportion of red blood cells in blood
  Day 4 | 0.0035 (0.00794)
  Day 7 | -0.0049 (0.01101)
  Day 10 | -0.0041 (0.01402)

23. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day -1) and at Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Trillion cells per liter | 0.170 (0.2080)

24. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 1 Day 9) and at Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Trillion cells per liter | 0.036 (0.1020)

25. Secondary Outcome: Period 3: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 2 Day 7) and at Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Trillion cells per liter
  Day 4 | 0.016 (0.0943)
  Day 7 | -0.079 (0.1038)
  Day 10 | -0.054 (0.1540)

26. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day -1) and at Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Femtoliter | 0.63 (0.774)

27. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 1 Day 9) and at Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Femtoliter | -0.86 (0.564)

28. Secondary Outcome: Period 3: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 2 Day 7) and at Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Femtoliter
  Day 4 | 0.40 (0.542)
  Day 7 | 0.36 (0.762)
  Day 10 | 0.05 (0.954)

29. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day -1) and at Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Picograms | -0.11 (0.279)

30. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 1 Day 9) and at Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Picograms | -0.17 (0.218)

31. Secondary Outcome: Period 3: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 2 Day 7) and at Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Picograms
  Day 4 | 0.55 (0.225)
  Day 7 | 0.55 (0.329)
  Day 10 | 0.52 (0.315)

32. Secondary Outcome: Period 1: Change From Baseline in Chemistry Parameters: Glucose, Cholesterol, Triglycerides, Anion Gap, Calcium, Carbon Dioxide, Chloride, Phosphate, Potassium, Sodium, Blood Urea Nitrogen
Description: Blood samples were collected to analyze the chemistry parameters: glucose, cholesterol, triglycerides, anion gap, calcium, carbon dioxide, chloride, phosphate, potassium, sodium and blood urea nitrogen. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day -1) and at Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Millimoles per liter
  Glucose | 0.063 (0.4235)
  Cholesterol | 0.088 (0.6858)
  Triglycerides | -0.084 (0.3983)
  Anion gap | -1.2 (1.33)
  Calcium | 0.025 (0.0599)
  Carbon dioxide | -0.1 (2.03)
  Chloride | 1.6 (2.63)
  Phosphate | 0.091 (0.1531)
  Potassium | 0.05 (0.356)
  Sodium | 0.3 (2.15)
  Blood urea nitrogen | 0.297 (0.9823)

33. Secondary Outcome: Period 2: Change From Baseline in Chemistry Parameters: Glucose, Cholesterol, Triglycerides, Anion Gap, Calcium, Carbon Dioxide, Chloride, Phosphate, Potassium, Sodium, Blood Urea Nitrogen
Description: Blood samples were collected to analyze the chemistry parameters: glucose, cholesterol, triglycerides, anion gap, calcium, carbon dioxide, chloride, phosphate, potassium, sodium and blood urea nitrogen. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 1 Day 9) and at Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Millimoles per liter
  Glucose | -0.249 (0.1748)
  Cholesterol | -0.269 (0.2363)
  Triglycerides | 0.087 (0.2374)
  Anion gap | 2.2 (1.52)
  Calcium | 0.014 (0.0245)
  Carbon dioxide | -1.3 (1.53)
  Chloride | -0.7 (1.78)
  Phosphate | 0.037 (0.0955)
  Potassium | -0.03 (0.272)
  Sodium | 0.3 (1.74)
  Blood urea nitrogen | -0.341 (0.3937)

34. Secondary Outcome: Period 3: Change From Baseline in Chemistry Parameters: Glucose, Cholesterol, Triglycerides, Anion Gap, Calcium, Carbon Dioxide, Chloride, Phosphate, Potassium, Sodium, Blood Urea Nitrogen
Description: Blood samples were collected to analyze the chemistry parameters: glucose, cholesterol, triglycerides, anion gap, calcium, carbon dioxide, chloride, phosphate, potassium, sodium and blood urea nitrogen. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 2 Day 7) and at Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Millimoles per liter
  Day 4: Glucose | 0.062 (0.1638)
  Day 7: Glucose | 0.103 (0.1806)
  Day 10: Glucose | -0.066 (0.2205)
  Day 4: Cholesterol | 0.096 (0.2400)
  Day 7: Cholesterol | -0.008 (0.2693)
  Day 10: Cholesterol | -0.030 (0.2366)
  Day 4: Triglycerides | 0.034 (0.2316)
  Day 7: Triglycerides | -0.094 (0.2578)
  Day 10: Triglycerides | 0.095 (0.2178)
  Day 4: Anion gap | -4.1 (1.24)
  Day 7: Anion gap | 0.1 (1.69)
  Day 10: Anion gap | 0.8 (1.65)
  Day 4: Calcium | -0.003 (0.0416)
  Day 7: Calcium | 0.026 (0.0413)
  Day 10: Calcium: | 0.035 (0.0561)
  Day 4: Carbon dioxide | 0.9 (1.65)
  Day 7: Carbon dioxide | 0.1 (1.59)
  Day 10: Carbon dioxide | 1.0 (2.16)
  Day 4: Chloride | 0.7 (1.92)
  Day 7: Chloride | -0.3 (1.39)
  Day 10: Chloride | -1.1 (1.86)
  Day 4: Phosphate | -0.004 (0.0808)
  Day 7: Phosphate | -0.013 (0.1151)
  Day 10: Phosphate | -0.051 (0.1115)
  Day 4: Potassium | -0.04 (0.239)
  Day 7: Potassium | -0.03 (0.218)
  Day 10: Potassium | 0.06 (0.189)
  Day 4: Sodium | -2.0 (1.37)
  Day 7: Sodium | -0.1 (1.65)
  Day 10: Sodium | 0.5 (1.90)
  Day 4: Blood urea nitrogen | 0.054 (0.5287)
  Day 7: Blood urea nitrogen | -0.178 (0.3542)
  Day 10: Blood urea nitrogen | -0.026 (0.5156)

35. Secondary Outcome: Period 1: Change From Baseline in Chemistry Parameters: Creatine Kinase, Lactate Dehydrogenase, Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Gamma-glutamyl Transferase
Description: Blood samples were collected to analyze the chemistry parameters: creatine kinase, lactate dehydrogenase, ALT, ALP, AST and gamma-glutamyl transferase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day -1) and at Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
International units per liter
  Creatine kinase | -32.0 (61.33)
  Lactate dehydrogenase | -21.9 (14.16)
  ALT | -0.3 (8.28)
  ALP | -0.1 (7.67)
  AST | -0.7 (3.36)
  Gamma-glutamyl transferase | -2.1 (3.13)

36. Secondary Outcome: Period 2: Change From Baseline in Chemistry Parameters: Creatine Kinase, Lactate Dehydrogenase, ALT, ALP, AST, Gamma-glutamyl Transferase
Description: Blood samples were collected to analyze the chemistry parameters: creatine kinase, lactate dehydrogenase, ALT, ALP, AST and gamma-glutamyl transferase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 1 Day 9) and at Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
International units per liter
  Creatine kinase | 22.6 (58.21)
  Lactate dehydrogenase | 9.1 (5.76)
  ALT | -0.6 (2.80)
  ALP | 1.9 (2.70)
  AST | 0.2 (1.87)
  Gamma-glutamyl transferase | -0.8 (1.28)

37. Secondary Outcome: Period 3: Change From Baseline in Chemistry Parameters: Creatine Kinase, Lactate Dehydrogenase, ALT, ALP, AST, Gamma-glutamyl Transferase
Description: Blood samples were collected to analyze the chemistry parameters: creatine kinase, lactate dehydrogenase, ALT, ALP, AST and gamma-glutamyl transferase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 2 Day 7) and at Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
International units per liter
  Day 4: Creatine kinase | -32.1 (131.30)
  Day 7: Creatine kinase | -37.1 (158.35)
  Day 10: Creatine kinase | -42.1 (162.94)
  Day 4: Lactate dehydrogenase | 5.9 (7.38)
  Day 7: Lactate dehydrogenase | -0.9 (7.02)
  Day 10: Lactate dehydrogenase | 0.1 (10.32)
  Day 4: ALT | 1.1 (4.36)
  Day 7: ALT | 0.7 (4.69)
  Day 10: ALT | 1.9 (4.11)
  Day 4: ALP | -1.6 (2.00)
  Day 7: ALP | -0.6 (2.39)
  Day 10: ALP | 0.8 (4.06)
  Day 4: AST | 0.9 (2.45)
  Day 7: AST | -0.5 (2.68)
  Day 10: AST | 0.3 (2.29)
  Day 4: Gamma-glutamyl transferase | -0.8 (0.75)
  Day 7: Gamma-glutamyl transferase | -0.3 (1.06)
  Day 10: Gamma-glutamyl transferase | 0.5 (1.51)

38. Secondary Outcome: Period 1: Change From Baseline in Chemistry Parameters: Urate, Creatinine, Bilirubin, Direct Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: urate, creatinine, bilirubin and direct bilirubin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day -1) and at Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Micromoles per liter
  Urate | -32.3 (42.01)
  Creatinine | 5.41 (7.253)
  Bilirubin | 0.01 (4.516)
  Direct bilirubin | 0.03 (0.677)

39. Secondary Outcome: Period 2: Change From Baseline in Chemistry Parameters: Urate, Creatinine, Bilirubin, Direct Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: urate, creatinine, bilirubin and direct bilirubin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 1 Day 9) and at Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Micromoles per liter
  Urate | -7.1 (14.52)
  Creatinine | -3.36 (4.219)
  Bilirubin | 0.27 (1.299)
  Direct bilirubin | 0.06 (0.328)

40. Secondary Outcome: Period 3: Change From Baseline in Chemistry Parameters: Urate, Creatinine, Bilirubin, Direct Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: urate, creatinine, bilirubin and direct bilirubin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 2 Day 7) and at Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Micromoles per liter
  Day 4: Urate | 0.0 (16.23)
  Day 7: Urate | -15.6 (26.39)
  Day 10: Urate | -1.4 (24.69)
  Day 4: Creatinine | 7.90 (4.239)
  Day 7: Creatinine | 9.89 (4.014)
  Day 10: Creatinine | 1.99 (4.739)
  Day 4: Bilirubin | 2.24 (2.659)
  Day 7: Bilirubin | -0.21 (1.455)
  Day 10: Bilirubin | 1.43 (2.011)
  Day 4: Direct bilirubin | 0.33 (0.425)
  Day 7: Direct bilirubin | -0.19 (0.436)
  Day 10: Direct bilirubin | 0.22 (0.248)

41. Secondary Outcome: Period 1: Change From Baseline in Chemistry Parameters: Albumin, Globulin, Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin, globulin and protein. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day -1) and at Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Grams per liter
  Albumin | 0.4 (2.45)
  Globulin | 0.8 (1.11)
  Protein | 1.2 (3.06)

42. Secondary Outcome: Period 2: Change From Baseline in Chemistry Parameters: Albumin, Globulin, Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin, globulin and protein. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 1 Day 9) and at Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Grams per liter
  Albumin | 0.9 (1.45)
  Globulin | -1.1 (0.77)
  Protein | -0.2 (1.76)

43. Secondary Outcome: Period 3: Change From Baseline in Chemistry Parameters: Albumin, Globulin, Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin, globulin and protein. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 2 Day 7) and at Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Grams per liter
  Day 4: Albumin | 0.9 (1.00)
  Day 7: Albumin | 0.2 (1.22)
  Day 10: Albumin | 0.4 (2.06)
  Day 4: Globulin | -0.9 (1.29)
  Day 7: Globulin | 1.0 (1.10)
  Day 10: Globulin | 0.5 (1.32)
  Day 4: Protein | 0.0 (1.75)
  Day 7: Protein | 1.2 (1.80)
  Day 10: Protein | 0.9 (2.90)

44. Secondary Outcome: Period 1: Change From Baseline in Chemistry Parameters: Amylase, Lipase
Description: Blood samples were collected to analyze the chemistry parameters: amylase and lipase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day -1) and at Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Units per liter
  Amylase | 3.1 (9.63)
  Lipase | -3.4 (8.97)

45. Secondary Outcome: Period 2: Change From Baseline in Chemistry Parameters: Amylase, Lipase
Description: Blood samples were collected to analyze the chemistry parameters: amylase and lipase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 1 Day 9) and at Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Units per liter
  Amylase | -2.8 (4.65)
  Lipase | -0.7 (3.79)

46. Secondary Outcome: Period 3: Change From Baseline in Chemistry Parameters: Amylase, Lipase
Description: Blood samples were collected to analyze the chemistry parameters: amylase and lipase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 2 Day 7) and at Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Units per liter
  Day 4: Amylase | -1.6 (3.18)
  Day 7: Amylase | 0.1 (4.25)
  Day 10: Amylase | -0.9 (6.08)
  Day 4: Lipase | 4.7 (6.10)
  Day 7: Lipase | -0.8 (4.76)
  Day 10: Lipase | 0.1 (5.24)

47. Secondary Outcome: Period 1: Change From Baseline in Urinalysis Parameter: Specific Gravity
Description: Urine samples were collected to analyze the urinalysis parameter: specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day -1) and at Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Ratio | 0.0053 (0.00865)

48. Secondary Outcome: Period 2: Change From Baseline in Urinalysis Parameter: Specific Gravity
Description: Urine samples were collected to analyze the urinalysis parameter: specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 1 Day 9) and at Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Ratio | -0.0004 (0.00645)

49. Secondary Outcome: Period 3: Change From Baseline in Urinalysis Parameter: Specific Gravity
Description: Urine samples were collected to analyze the urinalysis parameter: specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 2 Day 7) and at Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Ratio
  Day 4 | 0.0003 (0.00652)
  Day 7 | -0.0007 (0.00545)
  Day 10 | -0.0016 (0.00901)

50. Secondary Outcome: Period 1: Change From Baseline in Urinalysis Parameter: Urobilinogen
Description: Urine samples were collected to analyze the urinalysis parameter: urobilinogen. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day -1) and at Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Micromoles per liter | 0.0000 (0.00000)

51. Secondary Outcome: Period 2: Change From Baseline in Urinalysis Parameter: Urobilinogen
Description: Urine samples were collected to analyze the urinalysis parameter: urobilinogen. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 1 Day 9) and at Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Micromoles per liter | 0.0000 (0.00000)

52. Secondary Outcome: Period 3: Change From Baseline in Urinalysis Parameter: Urobilinogen
Description: Urine samples were collected to analyze the urinalysis parameter: urobilinogen. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 2 Day 7) and at Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Micromoles per liter
  Day 4 | 0.0000 (0.00000)
  Day 7 | 0.0000 (0.00000)
  Day 10 | 0.0000 (0.00000)

53. Secondary Outcome: Period 1: Change From Baseline in Urinalysis Parameter: Potential of Hydrogen (pH)
Description: Urine samples were collected to analyze the urinalysis parameter: pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day -1) and at Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
pH | -0.22 (0.730)

54. Secondary Outcome: Period 2: Change From Baseline in Urinalysis Parameter: pH
Description: Urine samples were collected to analyze the urinalysis parameter: pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 1 Day 9) and at Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
pH | 0.13 (0.428)

55. Secondary Outcome: Period 3: Change From Baseline in Urinalysis Parameter: pH
Description: Urine samples were collected to analyze the urinalysis parameter: pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first treatment in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Period 2 Day 7) and at Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
pH
  Day 4 | 0.03 (0.531)
  Day 7 | -0.13 (0.500)
  Day 10 | 0.16 (0.569)

56. Secondary Outcome: Period 1: Number of Participants With Urinalysis Dipstick Results
Description: Urine samples were collected at indicated time points to analyze parameters including glucose, protein, occult blood, ketones, nitrite, bilirubin and leukocyte esterase levels by dipstick. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters can be read as negative, Trace, 1+ (low concentrations present) and 2+ (moderate concentrations present) indicating proportional concentrations in the urine sample.
Time Frame: Day 9
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Participants
  Bilirubin: Negative | 16
  Glucose: Negative | 16
  Ketones: Negative | 15
  Ketones: Trace | 1
  Leukocyte Esterase: Negative | 16
  Nitrite: Negative | 16
  Occult Blood: Negative | 15
  Occult Blood: 2+ | 1
  Protein: Negative | 16

57. Secondary Outcome: Period 2: Number of Participants With Urinalysis Dipstick Results
Description: Urine samples were collected at indicated time points to analyze parameters including glucose, protein, occult blood, ketones, nitrite, bilirubin and leukocyte esterase levels by dipstick. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters can be read as negative, Trace, 1+ (low concentrations present), and 2+ (moderate concentrations present) indicating proportional concentrations in the urine sample.
Time Frame: Day 7
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Participants
  Bilirubin: Negative | 16
  Glucose: Negative | 16
  Ketones: Negative | 15
  Ketones: 1+ | 1
  Leukocyte Esterase: Negative | 15
  Leukocyte Esterase: 1+ | 1
  Nitrite: Negative | 16
  Occult Blood: Negative | 16
  Protein: Negative | 16

58. Secondary Outcome: Period 3: Number of Participants With Urinalysis Dipstick Results
Description: Urine samples were collected at indicated time points to analyze parameters including glucose, protein, occult blood, ketones, nitrite, bilirubin and leukocyte esterase levels by dipstick. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters can be read as negative, Trace, 1+ (low concentrations present), and 2+ (moderate concentrations present)indicating proportional concentrations in the urine sample.
Time Frame: Days 4, 7 and 10
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Participants
  Bilirubin: Day 4, Negative | 16
  Bilirubin: Day 7, Negative | 16
  Bilirubin: Day 10, Negative | 16
  Glucose: Day 4, Negative | 16
  Glucose: Day 7, Negative | 16
  Glucose: Day 10, Negative | 16
  Ketones: Day 4, Negative | 16
  Ketones: Day 7, Negative | 16
  Ketones: Day 10, Negative | 16
  Leukocyte Esterase: Day 4, Negative | 16
  Leukocyte Esterase: Day 7, Negative | 16
  Leukocyte Esterase: Day 10, Negative | 16
  Nitrite: Day 4, Negative | 16
  Nitrite: Day 7, Negative | 16
  Nitrite: Day 10, Negative | 16
  Occult Blood: Day 4, Negative | 16
  Occult Blood: Day 7, Negative | 16
  Occult Blood: Day 10, Negative | 16
  Protein: Day 4, Negative | 16
  Protein: Day 7, Negative | 16
  Protein: Day 10, Negative | 16

59. Secondary Outcome: Period 1: Change From Baseline in PR Interval, QRS Duration, QT Interval, Fridericia QT Correction Formula (QTcF), Bazett's QT Correction Formula (QTcB)
Description: Twelve-lead electrocardiograms (ECG) were obtained to measure PR Interval, QRS Duration, QT Interval, QTcF Interval and QTcB Interval. Twelve-lead ECGs were performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes. Baseline was defined as the average of the triplicate pre-dose assessments on Day 1 of Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline, Day 1: 2 hours, 4 hours; Day 5: Pre-dose, 2 hours and 4 hours
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Milliseconds
  PR Interval: Day 1, 2 hours | -0.5 (9.33)
  PR Interval: Day 1, 4 hours | 1.7 (8.34)
  PR Interval: Day 5, Pre-dose | 4.7 (6.32)
  PR Interval: Day 5, 2 hours | 1.3 (8.52)
  PR Interval: Day 5, 4 hours | 1.9 (12.94)
  QRS Duration: Day 1, 2 hours | 1.8 (3.04)
  QRS Duration: Day 1, 4 hours | 1.3 (3.32)
  QRS Duration: Day 5, Pre-dose | -0.8 (3.21)
  QRS Duration: Day 5, 2 hours | 0.8 (3.99)
  QRS Duration: Day 5, 4 hours | 0.6 (2.78)
  QT Interval: Day 1, 2 hours | -5.5 (8.21)
  QT Interval: Day 1, 4 hours | 9.9 (12.91)
  QT Interval: Day 5, Pre-dose | -6.8 (11.74)
  QT Interval: Day 5, 2 hours | -16.3 (16.64)
  QT Interval: Day 5, 4 hours | 1.2 (16.07)
  QTcF Interval: Day 1, 2 hours | -5.0 (8.42)
  QTcF Interval: Day 1, 4 hours | -1.6 (8.52)
  QTcF Interval: Day 5, Pre-dose | -7.1 (8.53)
  QTcF Interval: Day 5, 2 hours | -7.9 (9.92)
  QTcF Interval: Day 5, 4 hours | -3.9 (7.56)
  QTcB Interval: Day 1, 2 hours | -4.5 (10.26)
  QTcB Interval: Day 1, 4 hours | -7.4 (9.16)
  QTcB Interval: Day 5, Pre-dose | -6.7 (8.16)
  QTcB Interval: Day 5, 2 hours | -3.4 (10.84)
  QTcB Interval: Day 5, 4 hours | -5.9 (11.62)

60. Secondary Outcome: Period 2: Change From Baseline in PR Interval, QRS Duration, QT Interval, QTcF, QTcB
Description: Twelve-lead ECG were obtained to measure PR Interval, QRS Duration, QT Interval, QTcF Interval and QTcB Interval. Twelve-lead ECGs were performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes. Baseline was defined as the average of the triplicate pre-dose assessments on Day 1 of Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline; Day 1: 2 hours, 4 hours; Day 5: Pre-dose, 2 hours and 4 hours
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Milliseconds
  PR Interval: Day 1, 2 hours | -3.3 (6.31)
  PR Interval: Day 1, 4 hours | -3.0 (5.55)
  PR Interval: Day 5, Pre-dose | -2.1 (6.15)
  PR Interval: Day 5, 2 hours | -3.4 (7.81)
  PR Interval: Day 5, 4 hours | -6.4 (6.77)
  QRS Duration: Day 1, 2 hours | 0.1 (2.54)
  QRS Duration: Day 1, 4 hours | -1.1 (4.08)
  QRS Duration: Day 5, Pre-dose | 0.3 (3.89)
  QRS Duration: Day 5, 2 hours | -0.2 (3.85)
  QRS Duration: Day 5, 4 hours | 0.6 (2.70)
  QT Interval: Day 1, 2 hours | -7.9 (11.47)
  QT Interval: Day 1, 4 hours | 4.6 (13.48)
  QT Interval: Day 5, Pre-dose | 2.8 (17.38)
  QT Interval: Day 5, 2 hours | -7.1 (16.13)
  QT Interval: Day 5, 4 hours | 6.3 (20.51)
  QTcF Interval: Day 1, 2 hours | -1.3 (8.74)
  QTcF Interval: Day 1, 4 hours | 3.1 (6.44)
  QTcF Interval: Day 5, Pre-dose | 6.6 (6.79)
  QTcF Interval: Day 5, 2 hours | 3.7 (9.36)
  QTcF Interval: Day 5, 4 hours | 10.2 (10.44)
  QTcB Interval: Day 1, 2 hours | 2.4 (13.45)
  QTcB Interval: Day 1, 4 hours | 2.6 (12.62)
  QTcB Interval: Day 5, Pre-dose | 8.4 (5.92)
  QTcB Interval: Day 5, 2 hours | 9.9 (11.93)
  QTcB Interval: Day 5, 4 hours | 12.4 (8.57)

61. Secondary Outcome: Period 3: Change From Baseline in PR Interval, QRS Duration, QT Interval, QTcF, QTcB
Description: Twelve-lead ECG were obtained to measure PR Interval, QRS Duration, QT Interval, QTcF Interval and QTcB Interval. Twelve-lead ECGs were performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline; Day 1: 2 hours, 4 hours; Days 4, 5 and 7: Pre-dose, 2 hours and 4 hours; Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Milliseconds
  PR Interval: Day 1, 2 hours | 1.9 (7.47)
  PR Interval: Day 1, 4 hours | -1.9 (8.19)
  PR Interval: Day 4, Pre-dose | -0.4 (6.97)
  PR Interval: Day 4, 2 hours | 0.9 (8.48)
  PR Interval: Day 4, 4 hours | -2.9 (9.53)
  PR Interval: Day 5, Pre-dose | -1.4 (10.59)
  PR Interval: Day 5, 2 hours | -3.2 (9.13)
  PR Interval: Day 5, 4 hours | -2.7 (7.77)
  PR Interval: Day 7, Pre-dose | 3.6 (7.61)
  PR Interval: Day 7, 2 hours | -1.0 (9.47)
  PR Interval: Day 7, 4 hours | -0.4 (7.61)
  PR Interval: Day 10 | 2.3 (8.60)
  QRS Duration: Day 1, 2 hours | 1.1 (5.47)
  QRS Duration: Day 1, 4 hours | -2.1 (3.80)
  QRS Duration: Day 4, Pre-dose | 2.0 (5.61)
  QRS Duration: Day 4, 2 hours | -1.3 (3.09)
  QRS Duration: Day 4, 4 hours | 0.5 (6.63)
  QRS Duration: Day 5, Pre-dose | 1.8 (6.18)
  QRS Duration: Day 5, 2 hours | 1.3 (5.11)
  QRS Duration: Day 5, 4 hours | -0.5 (3.31)
  QRS Duration: Day 7, Pre-dose | 0.6 (3.58)
  QRS Duration: Day 7, 2 hours | 0.3 (4.93)
  QRS Duration: Day 7, 4 hours | -0.4 (3.72)
  QRS Duration: Day 10 | 1.7 (5.45)
  QT Interval: Day 1, 2 hours | -7.8 (8.68)
  QT Interval: Day 1, 4 hours | 4.4 (13.15)
  QT Interval: Day 4, Pre-dose | 1.4 (14.28)
  QT Interval: Day 4, 2 hours | -11.2 (14.53)
  QT Interval: Day 4, 4 hours | 7.4 (13.68)
  QT Interval: Day 5, Pre-dose | -1.4 (13.57)
  QT Interval: Day 5, 2 hours | -6.9 (10.65)
  QT Interval: Day 5, 4 hours | 3.9 (14.59)
  QT Interval: Day 7, Pre-dose | 3.2 (17.34)
  QT Interval: Day 7, 2 hours | -5.6 (14.01)
  QT Interval: Day 7, 4 hours | 8.0 (15.38)
  QT Interval: Day 10 | 5.1 (10.39)
  QTcF Interval: Day 1, 2 hours | -0.4 (5.63)
  QTcF Interval: Day 1, 4 hours | 6.6 (4.97)
  QTcF Interval: Day 4, Pre-dose | 2.7 (8.21)
  QTcF Interval: Day 4, 2 hours | -2.5 (8.41)
  QTcF Interval: Day 4, 4 hours | 8.1 (9.10)
  QTcF Interval: Day 5, Pre-dose | 6.1 (8.14)
  QTcF Interval: Day 5, 2 hours | 1.1 (9.42)
  QTcF Interval: Day 5, 4 hours | 8.6 (6.26)
  QTcF Interval: Day 7, Pre-dose | 2.0 (9.21)
  QTcF Interval: Day 7, 2 hours | 0.6 (7.46)
  QTcF Interval: Day 7, 4 hours | 3.6 (7.28)
  QTcF Interval: Day 10 | 1.6 (7.36)
  QTcB Interval: Day 1, 2 hours | 3.8 (9.50)
  QTcB Interval: Day 1, 4 hours | 7.4 (10.78)
  QTcB Interval: Day 4, Pre-dose | 3.8 (13.72)
  QTcB Interval: Day 4, 2 hours | -0.6 (17.78)
  QTcB Interval: Day 4, 4 hours | 8.6 (12.83)
  QTcB Interval: Day 5, Pre-dose | 10.6 (13.25)
  QTcB Interval: Day 5, 2 hours | 5.5 (12.47)
  QTcB Interval: Day 5, 4 hours | 11.3 (9.50)
  QTcB Interval: Day 7, Pre-dose | 2.1 (14.09)
  QTcB Interval: Day 7, 2 hours | 4.4 (14.43)
  QTcB Interval: Day 7, 4 hours | 1.4 (10.35)
  QTcB Interval: Day 10 | 0.2 (10.89)

62. Secondary Outcome: Period 1: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in the semi-recumbent position with a completely automated device. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 2, 3, 4 and 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Millimeters of mercury
  SBP: Day 2 | 3.5 (9.97)
  SBP: Day 3 | -0.4 (8.88)
  SBP: Day 4 | 3.7 (11.97)
  SBP: Day 5 | -6.2 (8.88)
  DBP: Day 2 | 4.3 (6.70)
  DBP: Day 3 | 0.9 (9.89)
  DBP: Day 4 | 2.3 (8.50)
  DBP: Day 5 | -2.6 (10.70)

63. Secondary Outcome: Period 2: Change From Baseline in SBP and DBP
Description: SBP and DBP were measured in the semi-recumbent position with a completely automated device. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 2, 3, 4, 5, 6 and 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Millimeters of mercury
  SBP: Day 2 | 1.7 (5.19)
  SBP: Day 3 | 1.3 (6.83)
  SBP: Day 4 | 3.0 (7.73)
  SBP: Day 5 | -0.5 (5.40)
  SBP: Day 6 | -0.1 (8.01)
  SBP: Day 7 | 0.6 (4.57)
  DBP: Day 2 | -0.4 (7.03)
  DBP: Day 3 | 1.1 (4.46)
  DBP: Day 4 | -0.4 (4.67)
  DBP: Day 5 | -1.3 (4.85)
  DBP: Day 6 | 0.3 (6.37)
  DBP: Day 7 | 0.4 (5.62)

64. Secondary Outcome: Period 3: Change From Baseline in SBP and DBP
Description: SBP and DBP were measured in the semi-recumbent position with a completely automated device. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 2, 3, 4, 5, 6, 7, 8, 9, 10 and 11
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Millimeters of mercury
  SBP: Day 2 | -0.1 (7.66)
  SBP: Day 3 | -3.4 (6.54)
  SBP: Day 4 | -3.3 (6.63)
  SBP: Day 5 | 3.6 (17.17)
  SBP: Day 6 | -1.4 (7.08)
  SBP: Day 7 | -2.1 (7.76)
  SBP: Day 8 | -2.0 (9.36)
  SBP: Day 9 | -2.3 (8.00)
  SBP: Day 10 | -4.3 (8.35)
  SBP: Day 11 | -3.4 (7.69)
  DBP: Day 2 | 1.3 (3.32)
  DBP: Day 3 | -0.1 (5.73)
  DBP: Day 4 | 1.2 (4.51)
  DBP: Day 5 | 6.7 (22.20)
  DBP: Day 6 | 1.4 (6.99)
  DBP: Day 7 | 2.9 (5.88)
  DBP: Day 8 | 1.8 (9.89)
  DBP: Day 9 | 2.1 (5.87)
  DBP: Day 10 | 2.3 (4.91)
  DBP: Day 11 | -0.1 (5.43)

65. Secondary Outcome: Period 1: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in the semi-recumbent position with a completely automated device. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 2, 3, 4 and 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Beats per minute
  Day 2 | -0.3 (4.30)
  Day 3 | -1.3 (4.63)
  Day 4 | 2.0 (8.46)
  Day 5 | -1.6 (5.08)

66. Secondary Outcome: Period 2: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in the semi-recumbent position with a completely automated device. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 2, 3, 4, 5, 6 and 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Beats per minute
  Day 2 | 3.9 (8.54)
  Day 3 | 5.4 (7.19)
  Day 4 | 4.8 (7.50)
  Day 5 | 4.2 (8.73)
  Day 6 | 3.8 (6.51)
  Day 7 | 2.7 (5.78)

67. Secondary Outcome: Period 3: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in the semi-recumbent position with a completely automated device. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 2, 3, 4, 5, 6, 7, 8, 9, 10 and 11
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Beats per minute
  Day 2 | 1.8 (5.65)
  Day 3 | 2.2 (6.88)
  Day 4 | 0.3 (7.63)
  Day 5 | 3.1 (7.79)
  Day 6 | 1.3 (6.97)
  Day 7 | -2.1 (5.94)
  Day 8 | 2.3 (9.34)
  Day 9 | -0.8 (7.90)
  Day 10 | -2.9 (5.34)
  Day 11 | 1.7 (10.56)

68. Secondary Outcome: Period 1: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured in the semi-recumbent position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 2, 3, 4 and 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Breaths per minute
  Day 2 | -0.9 (3.18)
  Day 3 | 0.3 (2.05)
  Day 4 | -1.5 (3.06)
  Day 5 | -0.8 (2.29)

69. Secondary Outcome: Period 2: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured in the semi-recumbent position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 2, 3, 4, 5, 6 and 7
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Breaths per minute
  Day 2, n=16 | -0.5 (2.58)
  Day 3, n=16 | 0.4 (3.03)
  Day 4, n=16 | -0.6 (3.07)
  Day 5, n=15: number analyzed (Participants) | 15
  Day 5, n=15 | 1.3 (2.47)
  Day 6, n=16 | -0.4 (2.55)
  Day 7, n=16 | 0.1 (3.30)

70. Secondary Outcome: Period 3: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured in the semi-recumbent position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 2, 3, 4, 5, 6, 7, 8, 9, 10 and 11
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Breaths per minute
  Day 2 | 1.4 (3.07)
  Day 3 | 0.5 (3.39)
  Day 4 | 0.3 (3.34)
  Day 5 | -0.5 (2.97)
  Day 6 | 0.6 (3.24)
  Day 7 | 0.3 (3.09)
  Day 8 | 1.4 (2.80)
  Day 9 | -0.4 (3.36)
  Day 10 | 1.4 (2.80)
  Day 11 | 2.8 (2.41)

71. Secondary Outcome: Period 1: Change From Baseline in Body Temperature
Description: Body temperature was measured in the semi-recumbent position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, in Period 1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 2, 3, 4 and 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Degrees Celsius
  Day 2 | -0.04 (0.326)
  Day 3 | -0.14 (0.287)
  Day 4 | -0.19 (0.370)
  Day 5 | 0.03 (0.275)

72. Secondary Outcome: Period 2: Change From Baseline in Body Temperature
Description: Body temperature was measured in the semi-recumbent position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, in Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 2, 3, 4, 5, 6 and 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Degrees Celsius
  Day 2 | -0.14 (0.299)
  Day 3 | -0.25 (0.415)
  Day 4 | -0.19 (0.294)
  Day 5 | -0.05 (0.363)
  Day 6 | -0.13 (0.300)
  Day 7 | -0.13 (0.373)

73. Secondary Outcome: Period 3: Change From Baseline in Body Temperature
Description: Body temperature was measured in the semi-recumbent position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, in Period 3. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 2, 3, 4, 5, 6, 7, 8, 9, 10 and 11
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Degrees Celsius
  Day 2 | -0.08 (0.286)
  Day 3 | -0.18 (0.423)
  Day 4 | 0.02 (0.229)
  Day 5 | 0.00 (0.175)
  Day 6 | -0.03 (0.318)
  Day 7 | 0.06 (0.287)
  Day 8 | -0.13 (0.458)
  Day 9 | -0.10 (0.329)
  Day 10 | -0.03 (0.291)
  Day 11 | 0.13 (0.302)

74. Secondary Outcome: Period 1: Absolute Values for Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelet Count
Description: Blood samples were collected to analyze the hematology parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelet count.
Time Frame: Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
10^9 cells per liter
  Basophils | 0.045 (0.0115)
  Eosinophils | 0.232 (0.1440)
  Lymphocytes | 2.023 (0.5931)
  Monocytes | 0.512 (0.1133)
  Neutrophils | 3.038 (0.7559)
  Platelet count | 270.2 (47.62)

75. Secondary Outcome: Period 2: Absolute Values for Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelet Count
Description: as for outcome 74
Time Frame: Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
10^9 cells per liter
  Basophils | 0.039 (0.0134)
  Eosinophils | 0.206 (0.0960)
  Lymphocytes | 1.869 (0.4383)
  Monocytes | 0.488 (0.1081)
  Neutrophils | 2.878 (0.6859)
  Platelet count | 264.2 (48.37)

76. Secondary Outcome: Period 3: Absolute Values for Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelet Count
Description: as for outcome 74
Time Frame: Days 4, 7 and 10
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
10^9 cells per liter
  Day 4: Basophils, n=16 | 0.043 (0.0165)
  Day 7: Basophils, n=16 | 0.046 (0.0196)
  Day 10: Basophils, n=16 | 0.042 (0.0142)
  Day 4: Eosinophils, n=16 | 0.206 (0.1120)
  Day 7: Eosinophils, n=16 | 0.211 (0.1512)
  Day 10: Eosinophils, n=16 | 0.171 (0.0874)
  Day 4: Lymphocytes, n=16 | 1.739 (0.3701)
  Day 7: Lymphocytes, n=16 | 1.837 (0.3916)
  Day 10: Lymphocytes, n=16 | 1.753 (0.3450)
  Day 4: Monocytes, n=16 | 0.537 (0.1821)
  Day 7: Monocytes, n=16 | 0.490 (0.1157)
  Day 10: Monocytes, n=16 | 0.470 (0.1128)
  Day 4: Neutrophils, n=16 | 3.321 (1.4579)
  Day 7: Neutrophils, n=16 | 2.954 (0.5600)
  Day 10: Neutrophils, n=16 | 3.082 (0.6649)
  Day 4: Platelet count, n=16 | 259.3 (46.03)
  Day 7: Platelet count, n=15: number analyzed (Participants) | 15
  Day 7: Platelet count, n=15 | 255.3 (46.20)
  Day 10: Platelet count, n=16 | 258.3 (42.92)

77. Secondary Outcome: Period 1: Absolute Values for Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin.
Time Frame: Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Grams per liter | 146.4 (8.02)

78. Secondary Outcome: Period 2: Absolute Values for Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin.
Time Frame: Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Grams per liter | 146.5 (8.68)

79. Secondary Outcome: Period 3: Absolute Values for Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin.
Time Frame: Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Grams per liter
  Day 4 | 149.8 (8.74)
  Day 7 | 147.1 (8.23)
  Day 10 | 147.7 (9.17)

80. Secondary Outcome: Period 1: Absolute Values for Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit.
Time Frame: Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Proportion of red blood cells in blood | 0.4419 (0.01697)

81. Secondary Outcome: Period 2: Absolute Values for Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit.
Time Frame: Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Proportion of red blood cells in blood | 0.4406 (0.01887)

82. Secondary Outcome: Period 3: Absolute Values for Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit.
Time Frame: Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Proportion of red blood cells in blood
  Day 4 | 0.4441 (0.01956)
  Day 7 | 0.4357 (0.01924)
  Day 10 | 0.4364 (0.02267)

83. Secondary Outcome: Period 1: Absolute Values for Hematology Parameter: Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes.
Time Frame: Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Trillion cells per liter | 5.143 (0.3580)

84. Secondary Outcome: Period 2: Absolute Values for Hematology Parameter: Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes.
Time Frame: Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Trillion cells per liter | 5.179 (0.3575)

85. Secondary Outcome: Period 3: Absolute Values for Hematology Parameter: Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes.
Time Frame: Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Trillion cells per liter
  Day 4 | 5.194 (0.3476)
  Day 7 | 5.099 (0.3798)
  Day 10 | 5.124 (0.3678)

86. Secondary Outcome: Period 1: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume.
Time Frame: Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Femtoliter | 86.22 (5.670)

87. Secondary Outcome: Period 2: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume.
Time Frame: Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Femtoliter | 85.36 (5.509)

88. Secondary Outcome: Period 3: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume.
Time Frame: Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Femtoliter
  Day 4 | 85.76 (5.323)
  Day 7 | 85.72 (5.117)
  Day 10 | 85.41 (5.030)

89. Secondary Outcome: Period 1: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin.
Time Frame: Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Picograms | 28.58 (2.446)

90. Secondary Outcome: Period 2: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin.
Time Frame: Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Picograms | 28.41 (2.385)

91. Secondary Outcome: Period 3: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin.
Time Frame: Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Picograms
  Day 4 | 28.96 (2.514)
  Day 7 | 28.96 (2.404)
  Day 10 | 28.93 (2.530)

92. Secondary Outcome: Period 1: Absolute Values for Chemistry Parameters: Glucose, Cholesterol, Triglycerides, Anion Gap, Calcium, Carbon Dioxide, Chloride, Phosphate, Potassium, Sodium, Blood Urea Nitrogen
Description: Blood samples were collected to analyze the chemistry parameters: glucose, cholesterol, triglycerides, anion gap, calcium, carbon dioxide, chloride, phosphate, potassium, sodium and blood urea nitrogen.
Time Frame: Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Millimoles per liter
  Glucose | 5.165 (0.4788)
  Cholesterol | 4.456 (0.6591)
  Triglycerides | 1.107 (0.5362)
  Anion gap | 9.2 (1.28)
  Calcium | 2.393 (0.0781)
  Carbon dioxide | 30.5 (1.15)
  Chloride | 103.8 (2.32)
  Phosphate | 1.244 (0.1658)
  Potassium | 4.31 (0.427)
  Sodium | 139.3 (2.52)
  Blood urea nitrogen | 5.406 (0.7575)

93. Secondary Outcome: Period 2: Absolute Values for Chemistry Parameters: Glucose, Cholesterol, Triglycerides, Anion Gap, Calcium, Carbon Dioxide, Chloride, Phosphate, Potassium, Sodium, Blood Urea Nitrogen
Description: as for outcome 92
Time Frame: Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Millimoles per liter
  Glucose | 4.916 (0.4825)
  Cholesterol | 4.187 (0.6783)
  Triglycerides | 1.194 (0.7294)
  Anion gap | 11.4 (1.20)
  Calcium | 2.406 (0.0772)
  Carbon dioxide | 29.3 (1.57)
  Chloride | 103.1 (2.35)
  Phosphate | 1.281 (0.1510)
  Potassium | 4.23 (0.249)
  Sodium | 139.6 (1.90)
  Blood urea nitrogen | 5.065 (0.6775)

94. Secondary Outcome: Period 3: Absolute Values for Chemistry Parameters: Glucose, Cholesterol, Triglycerides, Anion Gap, Calcium, Carbon Dioxide, Chloride, Phosphate, Potassium, Sodium, Blood Urea Nitrogen
Description: as for outcome 92
Time Frame: Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Millimoles per liter
  Day 4: Glucose | 4.978 (0.4655)
  Day 7: Glucose | 5.018 (0.3977)
  Day 10: Glucose | 4.849 (0.3858)
  Day 4: Cholesterol | 4.283 (0.8001)
  Day 7: Cholesterol | 4.179 (0.7438)
  Day 10: Cholesterol | 4.157 (0.8037)
  Day 4: Triglycerides | 1.228 (0.6403)
  Day 7: Triglycerides | 1.100 (0.5887)
  Day 10: Triglycerides | 1.289 (0.6625)
  Day 4: Anion gap | 7.3 (1.01)
  Day 7: Anion gap | 11.4 (1.75)
  Day 10: Anion gap | 12.1 (1.31)
  Day 4: Calcium | 2.404 (0.0855)
  Day 7: Calcium | 2.433 (0.0827)
  Day 10: Calcium | 2.441 (0.0681)
  Day 4: Carbon dioxide | 30.2 (1.56)
  Day 7: Carbon dioxide | 29.4 (1.15)
  Day 10: Carbon dioxide | 30.3 (1.53)
  Day 4: Chloride | 103.8 (2.77)
  Day 7: Chloride | 102.8 (2.07)
  Day 10: Chloride | 101.9 (2.02)
  Day 4: Phosphate | 1.276 (0.1304)
  Day 7: Phosphate | 1.268 (0.1802)
  Day 10: Phosphate | 1.229 (0.1213)
  Day 4: Potassium | 4.19 (0.150)
  Day 7: Potassium | 4.19 (0.217)
  Day 10: Potassium | 4.29 (0.275)
  Day 4: Sodium | 137.6 (2.06)
  Day 7: Sodium | 139.5 (2.56)
  Day 10: Sodium | 140.1 (2.11)
  Day 4: Blood urea nitrogen | 5.119 (0.8548)
  Day 7: Blood urea nitrogen | 4.887 (0.6388)
  Day 10: Blood urea nitrogen | 5.039 (0.8264)

95. Secondary Outcome: Period 1: Absolute Values for Chemistry Parameters: Creatine Kinase, Lactate Dehydrogenase, ALT, ALP, AST, Gamma-glutamyl Transferase
Description: Blood samples were collected to analyze the chemistry parameters: creatine kinase, lactate dehydrogenase, ALT, ALP, AST and gamma-glutamyl transferase.
Time Frame: Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
International units per liter
  Creatine kinase | 101.3 (57.10)
  Lactate dehydrogenase | 107.4 (14.33)
  ALT | 21.0 (10.71)
  ALP | 57.4 (8.74)
  AST | 16.6 (3.86)
  Gamma-glutamyl transferase | 21.1 (9.24)

96. Secondary Outcome: Period 2: Absolute Values for Chemistry Parameters: Creatine Kinase, Lactate Dehydrogenase, ALT, ALP, AST, Gamma-glutamyl Transferase
Description: as for outcome 95
Time Frame: Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
International units per liter
  Creatine kinase | 123.9 (112.28)
  Lactate dehydrogenase | 116.5 (15.10)
  ALT | 20.4 (9.88)
  ALP | 59.3 (9.19)
  AST | 16.8 (3.80)
  Gamma-glutamyl transferase | 20.3 (8.44)

97. Secondary Outcome: Period 3: Absolute Values for Chemistry Parameters: Creatine Kinase, Lactate Dehydrogenase, ALT, ALP, AST, Gamma-glutamyl Transferase
Description: as for outcome 95
Time Frame: Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
International units per liter
  Day 4: Creatine kinase | 110.3 (67.02)
  Day 7: Creatine kinase | 105.3 (63.83)
  Day 10: Creatine kinase | 100.3 (50.51)
  Day 4: Lactate dehydrogenase | 122.4 (16.26)
  Day 7: Lactate dehydrogenase | 115.6 (15.47)
  Day 10: Lactate dehydrogenase | 116.6 (18.79)
  Day 4: ALT | 21.4 (11.98)
  Day 7: ALT | 21.1 (12.00)
  Day 10: ALT | 22.3 (12.93)
  Day 4: ALP | 57.8 (9.34)
  Day 7: ALP | 58.8 (9.63)
  Day 10: ALP | 60.1 (9.07)
  Day 4: AST | 17.7 (5.12)
  Day 7: AST | 16.3 (4.78)
  Day 10: AST | 17.1 (4.55)
  Day 4: Gamma-glutamyl transferase | 19.5 (8.38)
  Day 7: Gamma-glutamyl transferase | 20.1 (8.35)
  Day 10: Gamma-glutamyl transferase | 20.8 (9.13)

98. Secondary Outcome: Period 1: Absolute Values for Chemistry Parameters: Urate, Creatinine, Bilirubin, Direct Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: urate, creatinine, bilirubin and direct bilirubin.
Time Frame: Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Micromoles per liter
  Urate | 321.9 (64.43)
  Creatinine | 90.28 (11.281)
  Bilirubin | 9.14 (2.423)
  Direct bilirubin | 1.87 (0.551)

99. Secondary Outcome: Period 2: Absolute Values for Chemistry Parameters: Urate, Creatinine, Bilirubin, Direct Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: urate, creatinine, bilirubin and direct bilirubin.
Time Frame: Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Micromoles per liter
  Urate | 314.8 (69.34)
  Creatinine | 86.92 (11.567)
  Bilirubin | 9.41 (3.014)
  Direct bilirubin | 1.93 (0.704)

100. Secondary Outcome: Period 3: Absolute Values for Chemistry Parameters: Urate, Creatinine, Bilirubin, Direct Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: urate, creatinine, bilirubin and direct bilirubin.
Time Frame: Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Micromoles per liter
  Day 4: Urate | 314.8 (65.44)
  Day 7: Urate | 299.3 (62.85)
  Day 10: Urate | 313.4 (60.33)
  Day 4: Creatinine | 94.82 (13.650)
  Day 7: Creatinine | 96.81 (12.861)
  Day 10: Creatinine | 88.91 (12.545)
  Day 4: Bilirubin | 11.64 (4.856)
  Day 7: Bilirubin | 9.19 (2.511)
  Day 10: Bilirubin | 10.83 (3.796)
  Day 4: Direct bilirubin | 2.26 (0.995)
  Day 7: Direct bilirubin | 1.74 (0.617)
  Day 10: Direct bilirubin | 2.15 (0.784)

101. Secondary Outcome: Period 1: Absolute Values for Chemistry Parameters: Albumin, Globulin, Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin, globulin and protein.
Time Frame: Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Grams per liter
  Albumin | 44.1 (3.32)
  Globulin | 27.9 (3.59)
  Protein | 71.9 (4.63)

102. Secondary Outcome: Period 2: Absolute Values for Chemistry Parameters: Albumin, Globulin, Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin, globulin and protein.
Time Frame: Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Grams per liter
  Albumin | 44.9 (3.13)
  Globulin | 26.8 (3.78)
  Protein | 71.8 (4.73)

103. Secondary Outcome: Period 3: Absolute Values for Chemistry Parameters: Albumin, Globulin, Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin, globulin and protein.
Time Frame: Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Grams per liter
  Day 4: Albumin | 45.9 (3.12)
  Day 7: Albumin | 45.1 (2.83)
  Day 10: Albumin | 45.3 (2.80)
  Day 4: Globulin | 25.9 (3.52)
  Day 7: Globulin | 27.8 (3.49)
  Day 10: Globulin | 27.3 (3.34)
  Day 4: Protein | 71.8 (3.89)
  Day 7: Protein | 72.9 (4.28)
  Day 10: Protein | 72.6 (4.11)

104. Secondary Outcome: Period 1: Absolute Values for Chemistry Parameters: Amylase, Lipase
Description: Blood samples were collected to analyze the chemistry parameters: amylase and lipase.
Time Frame: Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Units per liter
  Amylase | 59.6 (21.96)
  Lipase | 22.4 (8.57)

105. Secondary Outcome: Period 2: Absolute Values for Chemistry Parameters: Amylase, Lipase
Description: Blood samples were collected to analyze the chemistry parameters: amylase and lipase.
Time Frame: Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Units per liter
  Amylase | 56.8 (19.06)
  Lipase | 21.7 (7.34)

106. Secondary Outcome: Period 3: Absolute Values for Chemistry Parameters: Amylase, Lipase
Description: Blood samples were collected to analyze the chemistry parameters: amylase and lipase.
Time Frame: Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Units per liter
  Day 4: Amylase | 55.3 (18.81)
  Day 7: Amylase | 56.9 (21.03)
  Day 10: Amylase | 55.9 (20.57)
  Day 4: Lipase | 26.4 (11.10)
  Day 7: Lipase | 20.9 (9.12)
  Day 10: Lipase | 21.8 (9.25)

107. Secondary Outcome: Period 1: Absolute Values for Urinalysis Parameter: Specific Gravity
Description: Urine samples were collected to analyze the urinalysis parameter: specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine.
Time Frame: Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Ratio | 1.0181 (0.00662)

108. Secondary Outcome: Period 2: Absolute Values for Urinalysis Parameter: Specific Gravity
Description: as for outcome 107
Time Frame: Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Ratio | 1.0176 (0.00552)

109. Secondary Outcome: Period 3: Absolute Values for Urinalysis Parameter: Specific Gravity
Description: as for outcome 107
Time Frame: Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Ratio
  Day 4 | 1.0179 (0.00712)
  Day 7 | 1.0169 (0.00640)
  Day 10 | 1.0160 (0.00747)

110. Secondary Outcome: Period 1: Absolute Values for Urinalysis Parameter: Urobilinogen
Description: Urine samples were collected to analyze the urinalysis parameter: urobilinogen.
Time Frame: Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Micromoles per liter | 3.3860 (0.00000)

111. Secondary Outcome: Period 2: Absolute Values for Urinalysis Parameter: Urobilinogen
Description: Urine samples were collected to analyze the urinalysis parameter: urobilinogen.
Time Frame: Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Micromoles per liter | 3.3860 (0.00000)

112. Secondary Outcome: Period 3: Absolute Values for Urinalysis Parameter: Urobilinogen
Description: Urine samples were collected to analyze the urinalysis parameter: urobilinogen.
Time Frame: Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Micromoles per liter
  Day 4 | 3.3860 (0.00000)
  Day 7 | 3.3860 (0.00000)
  Day 10 | 3.3860 (0.00000)

113. Secondary Outcome: Period 1: Absolute Values for Urinalysis Parameter: pH
Description: Urine samples were collected to analyze the urinalysis parameter: pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0).
Time Frame: Day 9
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
pH | 5.88 (0.465)

114. Secondary Outcome: Period 2: Absolute Values for Urinalysis Parameter: pH
Description: as for outcome 113
Time Frame: Day 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
pH | 6.00 (0.548)

115. Secondary Outcome: Period 3: Absolute Values for Urinalysis Parameter: pH
Description: as for outcome 113
Time Frame: Days 4, 7 and 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
pH
  Day 4 | 6.03 (0.591)
  Day 7 | 5.88 (0.387)
  Day 10 | 6.16 (0.473)

116. Secondary Outcome: Period 1: Absolute Values for ECG Parameters: PR Interval, QRS Duration, QT Interval, QTcF, QTcB
Description: Twelve-lead ECG were obtained to measure PR Interval, QRS Duration, QT Interval, QTcF Interval and QTcB Interval. Twelve-lead ECGs were performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes.
Time Frame: Day 1: 2 hours, 4 hours; Day 5: Pre-dose, 2 hours and 4 hours
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Milliseconds
  PR Interval: Day 1, 2 hours | 159.1 (14.42)
  PR Interval: Day 1, 4 hours | 161.3 (16.51)
  PR Interval: Day 5, Pre-dose | 164.3 (14.87)
  PR Interval: Day 5, 2 hours | 160.9 (11.34)
  PR Interval: Day 5, 4 hours | 161.5 (12.66)
  QRS Duration: Day 1, 2 hours | 95.2 (9.59)
  QRS Duration: Day 1, 4 hours | 94.7 (10.90)
  QRS Duration: Day 5, Pre-dose | 92.6 (8.39)
  QRS Duration: Day 5, 2 hours | 94.2 (10.78)
  QRS Duration: Day 5, 4 hours | 94.0 (9.26)
  QT Interval: Day 1, 2 hours | 386.4 (16.06)
  QT Interval: Day 1, 4 hours | 401.8 (19.94)
  QT Interval: Day 5, Pre-dose | 385.1 (13.96)
  QT Interval: Day 5, 2 hours | 375.6 (11.46)
  QT Interval: Day 5, 4 hours | 393.1 (18.80)
  QTcF Interval: Day 1, 2 hours | 391.6 (11.37)
  QTcF Interval: Day 1, 4 hours | 395.0 (12.90)
  QTcF Interval: Day 5, Pre-dose | 389.5 (10.92)
  QTcF Interval: Day 5, 2 hours | 388.6 (14.47)
  QTcF Interval: Day 5, 4 hours | 392.7 (14.11)
  QTcB Interval: Day 1, 2 hours | 393.1 (15.31)
  QTcB Interval: Day 1, 4 hours | 390.2 (16.01)
  QTcB Interval: Day 5, Pre-dose | 390.9 (14.91)
  QTcB Interval: Day 5, 2 hours | 394.2 (21.59)
  QTcB Interval: Day 5, 4 hours | 391.7 (19.71)

117. Secondary Outcome: Period 2: Absolute Values for ECG Parameters: PR Interval, QRS Duration, QT Interval, QTcF, QTcB
Description: as for outcome 116
Time Frame: Day 1: 2 hours, 4 hours; Day 5: Pre-dose, 2 hours and 4 hours
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Milliseconds
  PR Interval: Day 1, 2 hours | 165.1 (15.46)
  PR Interval: Day 1, 4 hours | 165.4 (14.32)
  PR Interval: Day 5, Pre-dose | 166.3 (16.89)
  PR Interval: Day 5, 2 hours | 165.0 (19.90)
  PR Interval: Day 5, 4 hours | 162.0 (13.64)
  QRS Duration: Day 1, 2 hours | 94.1 (9.66)
  QRS Duration: Day 1, 4 hours | 92.9 (9.20)
  QRS Duration: Day 5, Pre-dose | 94.3 (10.12)
  QRS Duration: Day 5, 2 hours | 93.9 (9.00)
  QRS Duration: Day 5, 4 hours | 94.7 (8.51)
  QT Interval: Day 1, 2 hours | 381.8 (14.37)
  QT Interval: Day 1, 4 hours | 394.4 (19.18)
  QT Interval: Day 5, Pre-dose | 392.6 (23.20)
  QT Interval: Day 5, 2 hours | 382.6 (17.13)
  QT Interval: Day 5, 4 hours | 396.0 (21.45)
  QTcF Interval: Day 1, 2 hours | 390.0 (13.74)
  QTcF Interval: Day 1, 4 hours | 394.4 (12.38)
  QTcF Interval: Day 5, Pre-dose | 397.9 (14.64)
  QTcF Interval: Day 5, 2 hours | 395.0 (14.70)
  QTcF Interval: Day 5, 4 hours | 401.5 (12.66)
  QTcB Interval: Day 1, 2 hours | 393.3 (18.57)
  QTcB Interval: Day 1, 4 hours | 393.4 (18.53)
  QTcB Interval: Day 5, Pre-dose | 399.2 (16.61)
  QTcB Interval: Day 5, 2 hours | 400.7 (20.02)
  QTcB Interval: Day 5, 4 hours | 403.2 (13.41)

118. Secondary Outcome: Period 3: Absolute Values for ECG Parameters: PR Interval, QRS Duration, QT Interval, QTcF, QTcB
Description: as for outcome 116
Time Frame: Day 1: 2 hours, 4 hours; Days 4, 5 and 7: Pre-dose, 2 hours and 4 hours; Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Milliseconds
  PR Interval: Day 1, 2 hours | 167.9 (13.86)
  PR Interval: Day 1, 4 hours | 164.1 (15.12)
  PR Interval: Day 4, Pre-dose | 165.6 (16.02)
  PR Interval: Day 4, 2 hours | 166.9 (15.67)
  PR Interval: Day 4, 4 hours | 163.1 (15.13)
  PR Interval: Day 5, Pre-dose | 164.6 (18.30)
  PR Interval: Day 5, 2 hours | 162.8 (12.71)
  PR Interval: Day 5, 4 hours | 163.3 (14.96)
  PR Interval: Day 7, Pre-dose | 169.6 (17.47)
  PR Interval: Day 7, 2 hours | 165.0 (15.69)
  PR Interval: Day 7, 4 hours | 165.6 (15.00)
  PR Interval: Day 10 | 168.3 (17.14)
  QRS Duration: Day 1, 2 hours | 95.9 (10.49)
  QRS Duration: Day 1, 4 hours | 92.8 (8.76)
  QRS Duration: Day 4, Pre-dose | 96.8 (9.41)
  QRS Duration: Day 4, 2 hours | 93.5 (8.21)
  QRS Duration: Day 4, 4 hours | 95.3 (8.79)
  QRS Duration: Day 5, Pre-dose | 96.6 (9.77)
  QRS Duration: Day 5, 2 hours | 96.1 (11.66)
  QRS Duration: Day 5, 4 hours | 94.3 (9.56)
  QRS Duration: Day 7, Pre-dose | 95.4 (9.44)
  QRS Duration: Day 7, 2 hours | 95.1 (9.52)
  QRS Duration: Day 7, 4 hours | 94.4 (9.30)
  QRS Duration: Day 10 | 96.5 (9.14)
  QT Interval: Day 1, 2 hours | 380.0 (12.90)
  QT Interval: Day 1, 4 hours | 392.3 (16.39)
  QT Interval: Day 4, Pre-dose | 389.2 (18.65)
  QT Interval: Day 4, 2 hours | 376.6 (18.49)
  QT Interval: Day 4, 4 hours | 395.3 (17.89)
  QT Interval: Day 5, Pre-dose | 386.4 (18.49)
  QT Interval: Day 5, 2 hours | 380.9 (13.91)
  QT Interval: Day 5, 4 hours | 391.8 (20.53)
  QT Interval: Day 7, Pre-dose | 391.0 (21.99)
  QT Interval: Day 7, 2 hours | 382.3 (13.85)
  QT Interval: Day 7, 4 hours | 395.8 (20.94)
  QT Interval: Day 10 | 392.9 (14.54)
  QTcF Interval: Day 1, 2 hours | 392.7 (11.45)
  QTcF Interval: Day 1, 4 hours | 399.7 (10.37)
  QTcF Interval: Day 4, Pre-dose | 395.8 (13.94)
  QTcF Interval: Day 4, 2 hours | 390.6 (12.33)
  QTcF Interval: Day 4, 4 hours | 401.2 (13.55)
  QTcF Interval: Day 5, Pre-dose | 399.2 (14.92)
  QTcF Interval: Day 5, 2 hours | 394.3 (12.83)
  QTcF Interval: Day 5, 4 hours | 401.7 (11.91)
  QTcF Interval: Day 7, Pre-dose | 395.1 (12.91)
  QTcF Interval: Day 7, 2 hours | 393.7 (12.69)
  QTcF Interval: Day 7, 4 hours | 396.8 (13.47)
  QTcF Interval: Day 10 | 394.8 (13.08)
  QTcB Interval: Day 1, 2 hours | 398.4 (15.81)
  QTcB Interval: Day 1, 4 hours | 402.0 (15.46)
  QTcB Interval: Day 4, Pre-dose | 398.4 (17.82)
  QTcB Interval: Day 4, 2 hours | 394.0 (21.41)
  QTcB Interval: Day 4, 4 hours | 403.1 (17.67)
  QTcB Interval: Day 5, Pre-dose | 405.1 (23.00)
  QTcB Interval: Day 5, 2 hours | 400.1 (18.05)
  QTcB Interval: Day 5, 4 hours | 405.9 (16.27)
  QTcB Interval: Day 7, Pre-dose | 396.6 (17.50)
  QTcB Interval: Day 7, 2 hours | 398.9 (21.21)
  QTcB Interval: Day 7, 4 hours | 396.0 (18.10)
  QTcB Interval: Day 10 | 394.8 (18.39)

119. Secondary Outcome: Period 1: Absolute Values for SBP and DBP
Description: SBP and DBP were measured in the semi-recumbent position with a completely automated device.
Time Frame: Days 2, 3, 4 and 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Millimeters of mercury
  SBP: Day 2 | 118.8 (8.57)
  SBP: Day 3 | 114.9 (8.09)
  SBP: Day 4 | 119.0 (9.81)
  SBP: Day 5 | 109.1 (7.16)
  DBP: Day 2 | 76.1 (6.53)
  DBP: Day 3 | 72.7 (8.32)
  DBP: Day 4 | 74.1 (8.58)
  DBP: Day 5 | 69.2 (9.77)

120. Secondary Outcome: Period 2: Absolute Values for SBP and DBP
Description: SBP and DBP were measured in the semi-recumbent position with a completely automated device.
Time Frame: Days 2, 3, 4, 5, 6 and 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Millimeters of mercury
  SBP: Day 2 | 115.8 (7.15)
  SBP: Day 3 | 115.3 (7.57)
  SBP: Day 4 | 117.1 (8.74)
  SBP: Day 5 | 113.6 (7.35)
  SBP: Day 6 | 113.9 (8.29)
  SBP: Day 7 | 114.6 (5.73)
  DBP: Day 2 | 69.6 (8.50)
  DBP: Day 3 | 71.1 (7.65)
  DBP: Day 4 | 69.6 (5.24)
  DBP: Day 5 | 68.8 (6.49)
  DBP: Day 6 | 70.3 (7.02)
  DBP: Day 7 | 70.4 (6.65)

121. Secondary Outcome: Period 3: Absolute Values for SBP and DBP
Description: SBP and DBP were measured in the semi-recumbent position with a completely automated device.
Time Frame: Days 2, 3, 4, 5, 6, 7, 8, 9, 10 and 11
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Millimeters of mercury
  SBP: Day 2 | 115.8 (8.12)
  SBP: Day 3 | 112.5 (5.81)
  SBP: Day 4 | 112.6 (6.11)
  SBP: Day 5 | 119.4 (19.70)
  SBP: Day 6 | 114.4 (7.45)
  SBP: Day 7 | 113.8 (8.13)
  SBP: Day 8 | 113.9 (6.72)
  SBP: Day 9 | 113.6 (7.67)
  SBP: Day 10 | 111.6 (6.38)
  SBP: Day 11 | 112.4 (7.69)
  DBP: Day 2 | 69.0 (6.46)
  DBP: Day 3 | 67.7 (6.52)
  DBP: Day 4 | 68.9 (6.33)
  DBP: Day 5 | 74.4 (21.90)
  DBP: Day 6 | 69.2 (8.27)
  DBP: Day 7 | 70.6 (5.78)
  DBP: Day 8 | 69.5 (9.34)
  DBP: Day 9 | 69.8 (5.98)
  DBP: Day 10 | 70.0 (5.14)
  DBP: Day 11 | 67.7 (4.32)

122. Secondary Outcome: Period 1: Absolute Values for Pulse Rate
Description: Pulse rate was measured in the semi-recumbent position with a completely automated device.
Time Frame: Days 2, 3, 4 and 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Beats per minute
  Day 2 | 67.8 (8.47)
  Day 3 | 66.8 (6.68)
  Day 4 | 70.1 (10.57)
  Day 5 | 66.4 (8.21)

123. Secondary Outcome: Period 2: Absolute Values for Pulse Rate
Description: Pulse rate was measured in the semi-recumbent position with a completely automated device.
Time Frame: Days 2, 3, 4, 5, 6 and 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Beats per minute
  Day 2 | 68.3 (9.75)
  Day 3 | 69.7 (8.65)
  Day 4 | 69.1 (8.21)
  Day 5 | 68.5 (11.14)
  Day 6 | 68.1 (8.88)
  Day 7 | 67.0 (8.95)

124. Secondary Outcome: Period 3: Absolute Values for Pulse Rate
Description: Pulse rate was measured in the semi-recumbent position with a completely automated device.
Time Frame: Days 2, 3, 4, 5, 6, 7, 8, 9, 10 and 11
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Beats per minute
  Day 2 | 68.4 (9.79)
  Day 3 | 68.9 (8.63)
  Day 4 | 66.9 (9.26)
  Day 5 | 69.8 (10.57)
  Day 6 | 67.9 (10.12)
  Day 7 | 64.6 (8.02)
  Day 8 | 69.0 (12.02)
  Day 9 | 65.9 (10.12)
  Day 10 | 63.8 (8.53)
  Day 11 | 68.4 (12.27)

125. Secondary Outcome: Period 1: Absolute Values for Respiratory Rate
Description: Respiratory rate was measured in the semi-recumbent position after at least 5 minutes of rest for the participant in a quiet setting without distractions.
Time Frame: Days 2, 3, 4 and 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Breaths per minute
  Day 2 | 13.5 (1.37)
  Day 3 | 14.6 (2.16)
  Day 4 | 12.9 (1.78)
  Day 5 | 13.6 (2.22)

126. Secondary Outcome: Period 2: Absolute Values for Respiratory Rate
Description: as for outcome 125
Time Frame: Days 2, 3, 4, 5, 6 and 7
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Breaths per minute
  Day 2, n=16 | 13.6 (0.81)
  Day 3, n=16 | 14.5 (2.00)
  Day 4, n=16 | 13.5 (1.15)
  Day 5, n=15: number analyzed (Participants) | 15
  Day 5, n=15 | 15.3 (2.09)
  Day 6, n=16 | 13.8 (2.52)
  Day 7, n=16 | 14.3 (2.18)

127. Secondary Outcome: Period 3: Absolute Values for Respiratory Rate
Description: as for outcome 125
Time Frame: Days 2, 3, 4, 5, 6, 7, 8, 9, 10 and 11
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Breaths per minute
  Day 2 | 15.0 (2.42)
  Day 3 | 14.1 (1.54)
  Day 4 | 13.9 (2.96)
  Day 5 | 13.1 (1.45)
  Day 6 | 14.3 (2.05)
  Day 7 | 13.9 (1.86)
  Day 8 | 15.0 (1.03)
  Day 9 | 13.3 (3.00)
  Day 10 | 15.0 (1.79)
  Day 11 | 16.4 (1.31)

128. Secondary Outcome: Period 1: Absolute Values for Body Temperature
Description: Body temperature was measured in the semi-recumbent position after at least 5 minutes of rest for the participant in a quiet setting without distractions.
Time Frame: Days 2, 3, 4 and 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Degrees Celsius
  Day 2 | 36.36 (0.303)
  Day 3 | 36.26 (0.287)
  Day 4 | 36.21 (0.361)
  Day 5 | 36.43 (0.270)

129. Secondary Outcome: Period 2: Absolute Values for Body Temperature
Description: as for outcome 128
Time Frame: Days 2, 3, 4, 5, 6 and 7
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Degrees Celsius
  Day 2 | 36.26 (0.339)
  Day 3 | 36.15 (0.361)
  Day 4 | 36.21 (0.318)
  Day 5 | 36.35 (0.306)
  Day 6 | 36.28 (0.309)
  Day 7 | 36.28 (0.394)

130. Secondary Outcome: Period 3: Absolute Values for Body Temperature
Description: as for outcome 128
Time Frame: Days 2, 3, 4, 5, 6, 7, 8, 9, 10 and 11
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Degrees Celsius
  Day 2 | 36.33 (0.284)
  Day 3 | 36.22 (0.369)
  Day 4 | 36.42 (0.412)
  Day 5 | 36.40 (0.405)
  Day 6 | 36.37 (0.366)
  Day 7 | 36.46 (0.371)
  Day 8 | 36.28 (0.451)
  Day 9 | 36.30 (0.337)
  Day 10 | 36.37 (0.294)
  Day 11 | 36.53 (0.307)

131. Secondary Outcome: Period 2: Time of Maximum Observed Concentration (Tmax) of GSK3640254 for GSK3640254 Arm
Description: as for outcome 7
Time Frame: Day 7: Pre-dose, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Hours | 5.000 [3.50 to 8.00]

132. Secondary Outcome: Period 3: Tmax of GSK3640254 for Dolutegravir + GSK3640254 Arm
Description: as for outcome 7
Time Frame: Day 7: Pre-dose, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Hours | 5.000 [3.50 to 8.00]

133. Secondary Outcome: Period 2: Apparent Terminal Phase Half-life (T1/2) of GSK3640254 for GSK3640254 Arm
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of GSK3640254. The pharmacokinetic parameters were calculated by standard non-compartmental analysis. Data could not be determined due to limited sampling points after final dosing (during elimination phase). An accurate determination of GSK3640254 half-life would require sampling up to 3 times half-life (3 * approximately 24 hours). However sampling in Period 2 was performed up to only 24 hours post-dose.
Time Frame: Day 7: Pre-dose, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | GSK3640254 200 mg
Number analyzed (Participants) | 16
Hours | NA (NA) — Data could not be determined due to limited sampling points after final dosing (during elimination phase). An accurate determination of GSK3640254 half-life would require sampling up to 3 times half-life (3 * approximately 24 hours).

134. Secondary Outcome: Period 3: T1/2 of GSK3640254 for Dolutegravir + GSK3640254 Arm
Description: as for outcome 7
Time Frame: Day 7: Pre-dose, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Hours | 23.417 (15.0)

135. Secondary Outcome: Period 1: Tmax of Dolutegravir for Dolutegravir Arm
Description: as for outcome 2
Time Frame: Day 5: Pre-dose, 1, 1.5, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Hours | 3.000 [1.00 to 4.50]

136. Secondary Outcome: Period 3: Tmax of Dolutegravir for Dolutegravir + GSK3640254 Arm
Description: as for outcome 2
Time Frame: Day 7: Pre-dose, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Hours | 3.000 [1.00 to 4.50]

137. Secondary Outcome: Period 1: T1/2 of Dolutegravir for Dolutegravir Arm
Description: as for outcome 2
Time Frame: Day 5: Pre-dose, 1, 1.5, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Dolutegravir 50 mg
Number analyzed (Participants) | 16
Hours | 14.492 (11.8)

138. Secondary Outcome: Period 3: T1/2 of Dolutegravir for Dolutegravir + GSK3640254 Arm
Description: as for outcome 2
Time Frame: Day 7: Pre-dose, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Dolutegravir 50 mg + GSK3640254 200 mg
Number analyzed (Participants) | 16
Hours | 14.690 (12.1)

ADVERSE EVENTS:
Time Frame: Non-SAEs and SAEs were collected from start of the study treatment up to Day 27
Description: Safety Population consisted of all participants who received at least 1 dose of study medication.
Arm/Group | Dolutegravir 50 mg | GSK3640254 200 mg | Dolutegravir 50 mg + GSK3640254 200 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/16 | 3/16 | 2/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dolutegravir 50 mg (N=16) | GSK3640254 200 mg (N=16) | Dolutegravir 50 mg + GSK3640254 200 mg (N=16)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Medical device site dermatitis (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 1
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT03816696/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT03816696/SAP_001.pdf